CLINICAL TRIAL: NCT01486121
Title: S.O.S. Ventilation - Sedation Optimisation Strategy For Mechanical Ventilation In Intensive Care Unit Patients
Brief Title: Sedation Optimisation Strategy (S.O.S.) Ventilation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8667
Record Dates: First submitted 2011-11-10; First posted 2011-12-06 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Surgery; Critical Illness; Mechanical Ventilation Complication; Organ Dysfunction Syndrome; Intensive Care Unit Syndrome
Keywords: Surgery; Critical illness; Mechanical ventilation; Organ dysfunction syndrome; Intensive Care Units Sedation; Analgesia; Treatment protocol; Nursing protocol; Outcome; Pain; Neurological disorders; Delirium; Muscular weakness; Psychological disorders; Anxiety; Depression; Stress disorders; Post-Traumatic
MeSH Terms: conditions — Critical Illness; Agnosia; Pain; Nervous System Diseases; Delirium; Muscle Weakness; Mental Disorders; Anxiety Disorders; Depression; Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- S.O.S.-V (Other)
  Interventions: Other: Therapy strategy
- Standard (No Intervention)

INTERVENTIONS:
Other: Therapy strategy — Sedation & mechanical ventilation
  Arms: S.O.S.-V

SUMMARY:
Use of sedatives and analgesics is common in mechanically ventilated patients hospitalized in Intensive Care Unit (ICU). That is called " sedation " and aimed to reduce both pain and anxiety and also to allow an effective and atraumatic mechanical ventilation. However, sedation excess and ventilator support excess, both in duration and intensity, are associated with an excess morbidity. Patients usually are systematically sedated after having been intubated. Then, sedation is stopped first before ventilator support is weaning. Several studies shown that rationalized protocols of sedation and ventilation orderings had a beneficial impact on non surgical patients' outcome. Feasibility of these protocols in surgical patients is still unknown. Moreover, no study has evaluated an optimized paired strategy of sedation-ventilation based on the priority setting of ventilation. This priority setting of ventilation should increase patient's comfort in spite of increasing sedatives and analgesics dosing. An paired sedation-ventilation protocol optimized for both duration and intensity of these treatments could improve surgical patients' outcome in ICU.

DETAILED DESCRIPTION:
Intervention group:

* Continuous use of sedatives and analgesics (commonly called "sedation") will be stopped upon enrolment.
* Ventilator asynchrony in Volume assist Controlled Ventilation (VCV) will be treated by switching to Pressure Support Ventilation (PSV) or adjusting setting of VCV.
* Pain, anxiety and agitation will be treated by priority setting of the mechanical ventilator aimed to deliver the most comfortable ventilator support and secondly by adding analgesics and/or psychoactive drugs without inducing a coma state.- Persistent ventilator asynchrony or persistent agitation will be treated by 6-hours continuous sedation periods.
* Extubation will be performed according to criteria defined by the national consensus on mechanical ventilation weaning, which are based on a daily spontaneous breathing trial in the absence of any sedation.

Control group (standard practices):

* Continuous use of sedatives and analgesics (commonly called "sedation") will be daily stopped according to criteria defined by the national consensus on sedation for ICU patients.- During the period before the interruption of sedation, ventilator asynchrony in VCV will be treated by increasing the depth of sedation and then the dose of opioids.
* During the period before the interruption of sedation, pain, anxiety and agitation will be treated by a priority adjustment of sedation according to the nurse driven protocol recommended by the national consensus on sedation for ICU patients.- During the period after the interruption of sedation, ventilator asynchrony will be treated by switching to the PSV mode. In case of return to VCV, asynchrony will be treated by restart of sedation.
* During the period after the interruption of sedation, pain, anxiety and agitation will be treated as for the intervention group.
* Extubation will be performed according to criteria defined by the national consensus on mechanical ventilation weaning, which are based on a daily spontaneous breathing trial in the absence of any sedation.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated patient in assist control mode after a surgical procedure expected to be ventilated for 12-hours or more
* At least 1 organ dysfunction according to SOFA score
* Non paralyzed because of neuromuscular blocking agents
* Body temperature > or equal 36°CAge > or equal 18
* Surrogate decision maker's consent

Exclusion Criteria:

* Patients without any surgical procedure (medical patients)
* Continuous mechanical ventilation for 24-hours or longer
* Hospitalisation in ICU for 7-days or longer
* Severe ARDS (Acrasis study criteria, New England J Med 2011)
* Neurological injury
* Active toxicomania
* Reduction or cessation of active treatment
* Patient under tutelage
* Pregnancy
* No French health insurance
* Enrollment in another study on sedation or mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time to successful intubation | for 48 hours after intubation
  Time to successful intubation is defined as time from randomization to extubation (or tracheotomy mask) for 48 hours.

SECONDARY OUTCOMES:
Dose and duration of sedation | Day 0 to Days 28
  Dose and duration of sedation
Type and duration of mechanical ventilation | Day 0 to Days 28
  Type and duration of mechanical ventilation
Complications acquired in ICU | Days 28
  Complications acquired in ICU stress ulcers ileus infections delirium neuromuscular weakness pain
Length of stay in ICU and hospital | up to 6 months
  Length of stay in ICU and hospital
Mortality | up to 12 months
  ICU mortality, 3 months mortality and 12 months mortality
Quality of life, anxiety, depression, post-traumatic stress disorder 3 and 12 months after ICU discharge | up to 6 months
  Quality of life, anxiety, depression, post-traumatic stress disorder 3 and 12 months after ICU discharge
Incidence and duration of organ dysfunctions | Day 1 to Days 5
  Incidence and duration of organ dysfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Gerald GC Chanques, MD, PhD, Principal Investigator — UH, Montpellier
Locations (3):
- France (3):
  - Department of Anesthesiology & Critical Care, Estaing University Hospital, Clermont-Ferrand
  - Department of Anesthesiology & Critical Care, St Eloi University Hospital, Montpellier
  - Department of Anesthesiology & Critical Care, Caremeau University Hospita, Nîmes

REFERENCES:
- [Derived] Chanques G, Conseil M, Roger C, Constantin JM, Prades A, Carr J, Muller L, Jung B, Belafia F, Cisse M, Delay JM, de Jong A, Lefrant JY, Futier E, Mercier G, Molinari N, Jaber S; SOS-Ventilation study investigators. Immediate interruption of sedation compared with usual sedation care in critically ill postoperative patients (SOS-Ventilation): a randomised, parallel-group clinical trial. Lancet Respir Med. 2017 Oct;5(10):795-805. doi: 10.1016/S2213-2600(17)30304-1. Epub 2017 Sep 18. PMID 28935558